CLINICAL TRIAL: NCT02127502
Title: VENUS: Validation of Septic Gene ExpressioN Using SeptiCyte®
Brief Title: VENUS: Septic Gene Expression Using SeptiCyte
Acronym: VENUS
Status: Completed | Type: Observational
Sponsor: Immunexpress (Industry)
Collaborators: Intermountain Health Care, Inc. (Other); Johns Hopkins University (Other); Rush University Medical Center (Other); Northwell Health (Other); Loyola University (Other); Grady Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VENUS-1024931
Record Dates: First submitted 2014-04-17; First posted 2014-04-30 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Sepsis; Systemic Inflammatory Response Syndrome (SIRS)
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients sepsis suspected

SUMMARY:
The investigators seek to evaluate a new test for determining presence of infection/sepsis as compared to non-infection/systemic inflammatory response syndrome among critically ill patients within the first 24 hours of their being hospitalized in an intensive care unit (ICU) within the first 7 days of hospitalization. The primary purpose of the study is to validate SeptiCyte® Lab in this population as compared to: 1) the doctor's impression and 2) existing clinical parameters. The investigators also hope to assess how well a related, new blood test, SeptID® identifies different types of infection, as compared to cultures and other lab tests.

ELIGIBILITY:
Inclusion Criteria:

1. 18-89 years old on the day of ICU admission
2. SIRS present as defined by the presence of two or more of the following:

   * Temperature > 38°C or < 36°C
   * Heart Rate > 90 beat/min
   * Tachypnea > 20/min or PaCO2 < 32 mmHg
   * White Blood Cell count > 12 000/mm3 or < 4 000/mm3 or > 10% immature neutrophils (bands)

Exclusion Criteria:

1. Consent not provided
2. Age less than 18 or greater than 89 years old on the day of ICU admission
3. Not admitted to ICU
4. Clinical cultures or serologies not obtained
5. Subject has been admitted to study hospital (or transferring facility) for ≥ 24 hours
6. Elective cardiac surgery patients with an expected duration in ICU of less than 24 hours.
7. Patients on non-prophylactic antibiotics for more than 24 hours prior to ICU admission
8. Delay of >24 hours between trial enrollment and sample draw time
9. Ethnic/racial category has completed enrollment.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill subjects, admitted to an Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
SeptiCyte® Lab score | Subjects will be followed for the duration of their hospital stay, an expected average of 7 days.

SECONDARY OUTCOMES:
Comparison of SeptiCyte® Lab score to Leukocytosis, Bandemia, & procalcitonin | Subjects will be followed for the duration of their hospital stay, an expected average of 7 days.

OTHER OUTCOMES:
SeptID® results | Subjects will be followed for the duration of their hospital stay, an expected average of 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Russell R. Miller, MD, MPH, Principal Investigator — Intermountain Medical Center
Locations (6):
- United States (6):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Northwell Health, New Hyde Park, New York
  - Intermountain Medical Center, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopansri BK, Miller Iii RR, Burke JP, Levy M, Opal S, Rothman RE, D'Alessio FR, Sidhaye VK, Balk R, Greenberg JA, Yoder M, Patel GP, Gilbert E, Afshar M, Parada JP, Martin GS, Esper AM, Kempker JA, Narasimhan M, Tsegaye A, Hahn S, Mayo P, McHugh L, Rapisarda A, Sampson D, Brandon RA, Seldon TA, Yager TD, Brandon RB. Physician agreement on the diagnosis of sepsis in the intensive care unit: estimation of concordance and analysis of underlying factors in a multicenter cohort. J Intensive Care. 2019 Feb 21;7:13. doi: 10.1186/s40560-019-0368-2. eCollection 2019. PMID 30828456
- [Derived] Miller RR 3rd, Lopansri BK, Burke JP, Levy M, Opal S, Rothman RE, D'Alessio FR, Sidhaye VK, Aggarwal NR, Balk R, Greenberg JA, Yoder M, Patel G, Gilbert E, Afshar M, Parada JP, Martin GS, Esper AM, Kempker JA, Narasimhan M, Tsegaye A, Hahn S, Mayo P, van der Poll T, Schultz MJ, Scicluna BP, Klein Klouwenberg P, Rapisarda A, Seldon TA, McHugh LC, Yager TD, Cermelli S, Sampson D, Rothwell V, Newman R, Bhide S, Fox BA, Kirk JT, Navalkar K, Davis RF, Brandon RA, Brandon RB. Validation of a Host Response Assay, SeptiCyte LAB, for Discriminating Sepsis from Systemic Inflammatory Response Syndrome in the ICU. Am J Respir Crit Care Med. 2018 Oct 1;198(7):903-913. doi: 10.1164/rccm.201712-2472OC. PMID 29624409